CLINICAL TRIAL: NCT06358326
Title: Dry Needling in Patients With Carpal Tunnel Syndrome
Brief Title: Dry Needling and Rehabilitatin Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Karabuk-1
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Dry Needling; Carpal Tunnel Syndrome; Myofacial Pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Facial Pain | interventions — Dry Needling; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about their groups (training group or the control group) and they will be evaluated and trained at different places and times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): In addition to the exercise given to the control group, the treatment group will receive dry needling in the carpal tunnel area, 2 days a week for 3 weeks, for a total of 5 sessions.
  Interventions: Other: Dry needling
- Control Group (Active Comparator): The control group will be taught and asked to perform stretching, nerve mobilization and tendon-shifting exercises for 3 weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Dry needling — In addition to stretching, nerve mobilization and tendon gliding exercises, a total of 5 sessions of dry needling will be performed for fascial mobilization, 2 days a week for 3 weeks.
  Arms: Treatment Group
Other: Control group — The physiotherapist will teach stretching, neuromobilization and tendon shifting exercises and will be asked to do them regularly for 3 weeks.
  Arms: Control Group

SUMMARY:
Dry needling is used for myofascial release. However, its effectiveness in carpal tunnel syndrome (CTS) is not well known. It is thought that dry needling may also be an effective treatment for CTS by providing relaxation in the fascial tissue. Therefore, this study will examine the effects of dry needling treatment on pain, function, range of motion, proprioception and disability in patients with CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy in the society, which develops due to compression of the median nerve in the carpal tunnel. With the compression of the median nerve, a pain, numbness and tingling sensation spreading to the hand and wrist affects daily living activities and reduces the quality of life. Thickening and myofascial restriction in the carpal tunnel area also contribute to this situation. For this reason, various treatment methods have been developed for CTS, ranging from conservative treatment to surgery. Dry needling is also an alternative treatment method that can be used for CTS. Dry needling allows the fascial tissue to loosen and re-enter the healing process, leading to a decrease in pain and an increase in quality of life. However, its effectiveness in patients with CTS is unknown. This study aimed to examine the effectiveness of dry needling in patients with CTS.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study.
2. Being between the ages of 18-65.
3. Being diagnosed with mild or moderate stage CTS as a result of the electroneurophysiological test.

Exclusion Criteria:

1. Having additional neurological, rheumatological and orthopedic disorders.
2. Having had previous hand surgery.
3. Having an additional acute neck, shoulder, elbow and hand problem.
4. Having a BMI of 40 kg/m2 and above.
5. Being pregnant.
6. As a result of the electroneurophysiological test, the data related to the median nerve are at a severe level.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Pain severity | Baseline and 3 weeks post-intervention
  It will be evaluated with the Visual Analogue Scale. The scale ranges from 1 to 10 at 10 mm intervals. 0 indicates absence of pain and the highest value of 10 indicates extreme pain.
Wrist range of motion | Baseline and 3 weeks post-intervention
  Wrist flexion, extension, ulnar deviation and radial deviation joint range degrees will be measured using a universal goniometer.
Position sense | Baseline and 3 weeks post-intervention
  In the evaluation of joint position sense (proprioception), wrist extension, elbow flexion and shoulder flexion movements will be evaluated with an inclinometer. An increase in deviation from the target angle indicates a worsening of position sense.
Severity of symptoms | Baseline and 3 weeks post-intervention
  The patients' CTS-related symptom severity and functional status will be evaluated with the Boston Carpal Tunnel Syndrome Questionnaire. The severity of the patient's strain is scored between 1-5. Higher scores indicate greater disability.
Hands activity level | Baseline and 3 weeks post-intervention
  Duruöz hand index will be used to evaluate hand-related activity limitations. The survey yields a total score of 0-90, with a higher score indicating greater activity restriction.
Nerve cross-sectional area | Baseline and 3 weeks post-intervention
  With ultrasonography, the doctor will measure the median nerve cross-sectional area of the individual and the distance between the median nerve flexor retinaculum.

CONTACTS AND LOCATIONS:
Overall Officials: Fidan Yılmaz, MsC, Principal Investigator — Pursaklar State Hospital; Emime EMİRMAHMUTOĞLU, Bachelors, Principal Investigator — Pursaklar State Hospital; Banu Gökçen BAYDOĞAN TAN, MD, Study Director — Pursaklar State Hospital
Locations (1):
- Pursaklar State Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No